CLINICAL TRIAL: NCT01002911
Title: Phase III Pilot Study - A Simple Randomized Trial of Conventional Versus Multimodal Prevention of Arrhythmia Device Infection
Brief Title: Prevention of Arrhythmia Device Infection Trial (PADIT Pilot)
Acronym: PADIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PADIT
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Arrythmias
Keywords: Device procedure; pacemaker; ICD; antibiotics
MeSH Terms: interventions — Cefazolin; Bacitracin; Cephalexin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aggressive Antibiotic therapy (Experimental): Patients receive preoperative intravenous antibiotics, intracavitary antibiotics during surgery and postoperative antibiotics.
  Interventions: Drug: Cefazolin, Bacitracin, Cefalexin
- Conventional Antibiotic Therapy (Active Comparator): Preoperative intravenous antibiotics
  Interventions: Drug: Cefazolin

INTERVENTIONS:
Drug: Cefazolin, Bacitracin, Cefalexin — Single does of Cefazolin 1-2 g iv given over 60-120 minutes, 60-120 minutes prior to skin incision, Bacitracin wash, Cefalexin 250-500 mg TID
  Arms: Aggressive Antibiotic therapy
Drug: Cefazolin — Cefazolin 1-2 g iv given over 60-120 minutes, 60-120 minutes prior to skin incision
  Arms: Conventional Antibiotic Therapy

SUMMARY:
The goal of the pilot study is to compare conventional antibiotic therapy to an aggressive antibiotic therapy plan for the prevention of arrhythmia device infection in high-risk patients undergoing arrhythmia device procedures. All antibiotics are approved for use and readily available.

DETAILED DESCRIPTION:
Infection can occur after surgery for either a pacemaker or an implantable defibrillation and can have very serious consequences. These infections are common and can be seen in as many as 2-3% of high-risk patients. Doctors use antibiotics to prevent these infections, but we do not know how much or how often to give the antibiotics to get the best effect. It is not known whether additional antibiotics during and after the operation would further reduce the risk of infection. This research study will compare two different ways of using common antibiotics to prevent infection during and following a device procedure. One way is the standard approach of a single dose before surgery and the other way uses more antibiotics. We do not know if either way is better. The purpose of this study therefore, is to compare two types of antibiotic therapy plans to better understand if one is most effective in preventing infection.

This study will provide the ability to evaluate the feasibility (i.e. site activation, enrollment, compliance, drop-out) and generate proof of concept for the larger clinical trial of 12,000 patients in all 25 Canadian Hospitals implanting ICDs, which will be submitted to the CIHR. Additionally, the study supports the continued initiatives of the network of physician investigators (Canadian Heart Rhythm Society Device Advisory Committee - CHRS DAC) collaborating to address arrhythmia procedures related clinical trials that will answer simple clinical questions that will focus initially on safety issues.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* One of the following planned device procedures:

  * ICD, pacemaker, CRT-P, CRT-D generator and/or lead replacement or
  * Pocket or lead revision or
  * System upgrade (insertion or attempted insertion of leads) or
  * New cardiac resynchronization therapy device implant (pacemaker or ICD)

Exclusion Criteria:

* Unable or unwilling to provide written informed consent
* Unable or unwilling to complete the study follow-up schedule
* Life expectancy < 12 months as per the opinion if the local investigator
* Allergy to or unable to tolerate cefazolin or clindamycin or vancomycin
* Allergy to or unable to tolerate intracavitary bacitracin or gentamicin or cefazolin
* Previously enrolled in this trial
* In another study that would confound the results of this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2009-12; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Hospitalization attributed to device infection. | Patients will have one follow-up visit at 12 months or earlier should a primary outcome event occur.

SECONDARY OUTCOMES:
1. Any treatment with antibiotics for suspected device infection. | Patients will have one follow-up visit at 12 months
2. Antibiotic therapy related adverse event. | Patients will have one follow-up visit at 12 months
3. Prolongation of hospitalization due to proven or suspected adverse events from the hospitalization. | Patients will have one follow-up visit at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Andrew Krahn, Principal Investigator — University of British Columbia
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Quebec, Ste-Foy, Quebec, Canada

REFERENCES:
- [Derived] Longtin Y, Gervais P, Birnie DH, Wang J, Alings M, Philippon F, Parkash R, Manlucu J, Angaran P, Rinne C, Coutu B, Low RA, Essebag V, Morillo C, Redfearn D, Toal S, Becker G, Degrace M, Thibault B, Crystal E, Tung S, LeMaitre J, Sultan O, Bennett M, Bashir J, Ayala-Paredes F, Rioux L, Hemels MEW, Bouwels LHR, Exner DV, Dorian P, Connolly SJ, Krahn AD. Impact of Choice of Prophylaxis on the Microbiology of Cardiac Implantable Electronic Device Infections: Insights From the Prevention of Arrhythmia Device Infection Trial (PADIT). Open Forum Infect Dis. 2021 Oct 14;8(11):ofab513. doi: 10.1093/ofid/ofab513. eCollection 2021 Nov. PMID 34859113
- [Derived] Birnie DH, Wang J, Alings M, Philippon F, Parkash R, Manlucu J, Angaran P, Rinne C, Coutu B, Low RA, Essebag V, Morillo C, Redfearn D, Toal S, Becker G, Degrace M, Thibault B, Crystal E, Tung S, LeMaitre J, Sultan O, Bennett M, Bashir J, Ayala-Paredes F, Gervais P, Rioux L, Hemels MEW, Bouwels LHR, Exner DV, Dorian P, Connolly SJ, Longtin Y, Krahn AD. Risk Factors for Infections Involving Cardiac Implanted Electronic Devices. J Am Coll Cardiol. 2019 Dec 10;74(23):2845-2854. doi: 10.1016/j.jacc.2019.09.060. PMID 31806127
- [Derived] Krahn AD, Longtin Y, Philippon F, Birnie DH, Manlucu J, Angaran P, Rinne C, Coutu B, Low RA, Essebag V, Morillo C, Redfearn D, Toal S, Becker G, Degrace M, Thibault B, Crystal E, Tung S, LeMaitre J, Sultan O, Bennett M, Bashir J, Ayala-Paredes F, Gervais P, Rioux L, Hemels MEW, Bouwels LHR, van Vlies B, Wang J, Exner DV, Dorian P, Parkash R, Alings M, Connolly SJ. Prevention of Arrhythmia Device Infection Trial: The PADIT Trial. J Am Coll Cardiol. 2018 Dec 18;72(24):3098-3109. doi: 10.1016/j.jacc.2018.09.068. PMID 30545448